CLINICAL TRIAL: NCT05395013
Title: Efficacy and Safety of Plastic, Covered and Uncovered Self-expandable Metal Stents in the Treatment of Malignant Biliary Obstructions (NEOSTENT)
Acronym: NEOSTENT
Status: Completed | Type: Observational
Sponsor: Azienda Unità Sanitaria Locale della Romagna (Other)
Responsible Party: Principal Investigator, Carlo Fabbri, Chief of Gastroenterology and Digestive Endoscopy Unit, Forlì-Cesena Hospitals, Azienda Unità Sanitaria Locale della Romagna
Other Study IDs: 3196
Record Dates: First submitted 2021-11-13; First posted 2022-05-27 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Common Bile Duct Stricture; Jaundice; Malignant
Keywords: Biliary Stent; Jaundice; Pancreatic cancer; Common bile duct cancer
MeSH Terms: conditions — Jaundice; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to evaluate the efficacy and safety of the various types of stents available for biliary drainage in patients with neoplastic stenosis of the common bile duct and to evaluate the adherence to the current guidelines available.

DETAILED DESCRIPTION:
Biliary drainage before surgery or chemotherapy is a common practice in patients with neoplastic stenosis of the common bile duct, often required by the presence of clinical conditions such as the onset of cholangitis or severe jaundice.

The endoscopic approach has now been identified by the literature as the preferential drainage route, due to a lower incidence of adverse effects, liver or intraperitoneal metastases and lower costs associated with this technique compared to percutaneous drainage.

The latest guidelines from the European Society of Gastrointestinal Endoscopy recommend the placement of a 10 mm diameter self-expandable metal stent (SEMS) as the first choice for endoscopic drainage in patients with extra-hepatic biliary stenosis of neoplastic origin. Compared to plastic stents, SEMS placement is associated with a lower risk of developing stent dysfunction and/or cholangitis, lower risk of reintervention, and better patient survival.

However, among the various types of metal stents available, to date there is no agreement on which type is the most suitable, as data on efficacy and post-interventional morbidity and mortality of the fully or partially covered and uncovered metal stents are contradictory.

The aim of the study is to evaluate the efficacy and safety of the various types of stents available for biliary drainage in patients with neoplastic stenosis of the common bile duct and to evaluate the adherence to the current guidelines available.

ELIGIBILITY:
Inclusion Criteria:

* Common bile duct stricture (i.e. jaundice and/or cholangitis) of malignant origin
* Patients > 18 years old
* Obtaining informed consent

Exclusion Criteria:

- Lack of sufficient clinical and laboratory data to define clinical efficacy and/or follow-up available <1 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with common bile duct stricture (i.e. jaundice and/or cholangitis) of malignant origin who underwent endoscopic drainage
Sampling Method: Non-Probability Sample
Enrollment: 3149 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Bilirubin decrease | From 2017 to 2021
  Rate of resolution of obstructive jaundice in short and long term (i.e. maintenance of patency and/or the need for reintervention) of the different types of biliary stent placed in patients with neoplastic stenosis of the common bile duct

SECONDARY OUTCOMES:
Rate of adverse events | From 2017 to 2021
  Rate of periprocedural complications (i.e. bleeding, pancreatitis, cholecystitis) after biliary stent placement
Rate of endoscopic reintervention | From 2017 to 2021
  Rate of stent disfunction requiring an additional endoscopic procedure
Rate of biliary cannulation and successful stent placement | From 2017 to 2021
  Rate of biliary cannulation and successful stent placement

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Morgagni-Pierantoni, Forlì, Forlì-Cesena, Italy